CLINICAL TRIAL: NCT04568304
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Study to Evaluate the Efficacy and Safety of Toripalimab Injection (JS001) in Combination With Standard Chemotherapy Versus Placebo in Combination With Standard Chemotherapy as the 1st-line Therapy for Treatment-naive Subjects With PD-L1-positive Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Study Evaluating Toripalimab Injection Combined With Standard Chemotherapy as a First-line Treatment for Locally Advanced or Metastatic Urothelial Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-038-III-UBC
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — toripalimab; Gemcitabine; Injections; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab Injection + chemotherapy group (Experimental)
  Interventions: Biological: Toripalimab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin for Injection / Carboplatin Injection
- Placebo + chemotherapy group (Placebo Comparator)
  Interventions: Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin for Injection / Carboplatin Injection; Drug: Placebo

INTERVENTIONS:
Biological: Toripalimab Injection — Toripalimab Injection 240 mg iv infusion on Day 1 of each 3-week cycle. The cumulative duration of Toripalimab Injection is up to 2 years.
  Arms: Toripalimab Injection + chemotherapy group
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine 1000mg/㎡ iv infusion, on Day 1 and Day 8 of each cycle, each treatment cycle is 3 weeks.
  The chemotherapy regimen will be administered for 6 cycles.
Drug: Cisplatin for Injection / Carboplatin Injection — Cisplatin 70mg/㎡ iv infusion, on Day 1 or Day 2 of each cycle, each treatment cycle is 3 weeks.
  Carboplatin AUC 4.5 iv infusion, on Day 1 or Day 2 of each cycle, each treatment cycle is 3 weeks.
  The chemotherapy regimen will be administered for 6 cycles.
Drug: Placebo — Placebo iv infusion on Day 1 of each 3-week cycle. The cumulative duration of placebo is up to 2 years.
  Arms: Placebo + chemotherapy group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of Toripalimab Injection in combination with chemotherapy compared to placebo in combination with chemotherapy in subjects with PD-L1-positive unresectable locally advanced or metastatic urothelial carcinoma who have received no previous systemic therapy.

ELIGIBILITY:
Inclusion criteria

1. Have full knowledge on this study and are willing to sign informed consent form (ICF);
2. Age 18-75 years at time of signing ICF, male or female;
3. The investigator judged that the subject is eligible for platinum-based chemotherapy;
4. Presence of histopathologically confirmed unresectable locally advanced (T4, any N; or any T, N2-3) or metastatic urothelial carcinoma;
5. No prior systemic anti-tumor therapy;
6. Subjects who are able to provide tumor tissue slides (≥ 5 slides) for PD-L1 test and the corresponding pathology report and whose PD-L1 test must be positive before randomization;
7. With at least one measurable lesion as per RECIST 1.1 criteria;
8. ECOG performance status score of 0-1;
9. Adequate function of vital organs.

Exclusion criteria

1. Have received anti-tumor treatments, including chemotherapy, radiotherapy or investigational product within 28 days before randomization;
2. Have received traditional Chinese medicines with anti-tumor activity or immunomodulators (eg. Interferon and Interleukin) within 14 days before randomization;
3. Previous use of anti-PD-1/PD-L1 agent or a drug acting on another co-inhibitory T cell receptor;
4. Subjects who are currently participating in or have participated in a study with investigational product within 4 weeks before administration;
5. Having received systemic corticosteroid therapy (dose equivalent to prednisone > 10 mg/day) within 14 days before randomization;
6. Subjects with active central nervous system (CNS) metastasis;
7. Grade 2 or higher peripheral neuropathy or hearing loss.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression-free survival (INV-PFS) as per RECIST 1.1 criteria | Approximately 3 years
  To evaluate the investigator-assessed progression-free survival following Toripalimab Injection in combination with chemotherapy compared to placebo in combination with chemotherapy in subjects with PD-L1-positive unresectable locally advanced or metastatic urothelial carcinoma who have received no previous systemic therapy

SECONDARY OUTCOMES:
IRC-PFS | Approximately 3 years
  Independent central radiological review committee-assessed progression-free survival as per RECIST1.1 criteria
INV-ORR, IRC-ORR | Approximately 3 years
  Investigator- and IRC-assessed overall response rate
INV-DCR, IRC-DCR | Approximately 3 years
  Investigator- and IRC-assessed disease control rate
INV-DoR, IRC- DoR | Approximately 3 years
  Investigator- and IRC-assessed duration of response
OS | Approximately 5 years
  Overall survival
OS rate at 1 year | Approximately 3 years
  Overall survival rate at 1 year
OS rate at 2 years | Approximately 4 years
  Overall survival rate at 2 years
INV-PFS rate and IRC-PFS rate at 6 months | Approximately 2.5 years
  Investigator- and IRC-assessed progression-free survival rate at 6 months
INV-PFS rate and IRC-PFS rate at 1 year | Approximately 3 years
  Investigator- and IRC-assessed progression-free survival rate at 1 year
Incidence of AEs/SAEs | Approximately 4 years
  Study drug related adverse events, serious adverse events graded in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0

OTHER OUTCOMES:
Investigator-assessed PFS | Approximately 4 years
  Investigator-assessed progression-free survival to explore the efficacy of crossover to Toripalimab Injection in control group
Investigator-assessed ORR | Approximately 4 years
  Investigator-assessed overall response rate to explore the efficacy of crossover to Toripalimab Injection in control group
Investigator-assessed DCR | Approximately 4 years
  Investigator-assessed disease control rate to explore the efficacy of crossover to Toripalimab Injection in control group
Investigator-assessed DoR | Approximately 4 years
  Investigator-assessed duration of response to explore the efficacy of crossover to Toripalimab Injection in control group

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University Cancer Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai